CLINICAL TRIAL: NCT07221422
Title: The PREGNANT (Pregnant Resident Empowerment, GuidaNce, and Advocacy iN Training) Coaching Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erika Rangel, MD, Associate Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025P000907
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Burnout, Professional; Well-Being, Psychological; Imposter Phenomenon; Self Efficacy; Quality of Life
MeSH Terms: conditions — Burnout, Professional; Psychological Well-Being; imposter syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention participants will not be given protected time to participate and will have the same clinical workload as controls. They will meet monthly with a novice physician coach of their choice (one-on-one) and a certified physician coach (with an assigned group of 6 peers). To build community, participants are encouraged to attend sessions with their coaching group, but we will accommodate full schedules by allowing (1) participation in sessions with other coaching groups, (2) asynchronous video learning including self-guided exercises. Video conferencing will be used to facilitate attendance and scalability.
  Interventions: Behavioral: Coaching Program
- Control (Other): Delayed intervention. At the conclusion of the study, control participants will be offered a 2-hour workshop (led by a certified coach) covering group session topics, provided access to the videos, and given self-guided exercises used for asynchronous learning.
  Interventions: Behavioral: Coaching Program

INTERVENTIONS:
Behavioral: Coaching Program — Novel, 4-month coaching program tailored to the childbearing trainees. This consists of 4 1:1 coaching sessions with a novice faculty coach and 4 group sessions with a certified coach.

SUMMARY:
This is a mixed-methods study designed to develop and evaluate an innovative coaching program for physician trainee mothers. Approximately 48 participants will be recruited from informational flyers posted in resident work areas and distributed by program directors and GME. Interested participants will email study staff. Participants will be randomized to the control or intervention arm. Intervention participants will meet monthly with a novice physician coach of their choice (one-on-one) and a certified physician coach (with an assigned group of 6 peers through video-conferencing).

Participants in both arms of the study will respond to surveys at three points: enrollment (baseline), 4 months, and 7 months. At each point, they will spend approximately 10 minutes filling the survey. The survey will query demographics, burnout, professional fulfillment, imposter phenomenon, self-valuation, self-efficacy, resilience, quality of life, and impact of work on professional relationships. The coaching intervention will last 4 months, and the 7 month survey will be used only to assess long-term effects of the intervention. At the conclusion of the study (7 months after enrollment), participants will be interviewed over video communication (secure Partners or Harvard Zoom) for approximately 30 minutes.

DETAILED DESCRIPTION:
To bridge the gaps identified in traditional mentorship programs, the PREGNANT study aims to develop and evaluate a novel, 4-month coaching program tailored to the childbearing trainees. Professional coaching is one of the few interventions shown to be effective in reducing burnout by providing structured and unstructured discussions through active listening and goal setting. It is uniquely positioned to address gaps identified in the previous mentorship program, as it does not rely on shared experiences, offers a focused solution with clear objectives, and provides trainees the tools to sustainably reduce burnout by fostering resilience, self-efficacy, and self-compassion. Despite its efficacy, many coaching programs rely on resource-intensive, in-person interventions, which reduce accessibility for trainees and pose scalability challenges.To overcome these barriers, our pilot study draws on the success of two types of innovative programs: 1) those that increase number of available one-on-one coaches by training practicing physicians in coaching techniques so they can function as "novice coaches" and 2) web-based group coaching programs with asynchronous learning opportunities, led by certified physician coaches, ensuring accessibility for trainees regardless of geographical or scheduling constraints. Unlike traditional life-coaching interventions that use external non-physician consultants, this program will be delivered by physician coaches who understand the challenges, social hierarchy, and culture of medical training. This distinction ensures that coaching is relevant and contextualized to the realities faced by childbearing trainees, thereby enhancing its effectiveness and impact.

This initiative will purposively include lesbian, gay, bisexual, transgender, queer, and other sexual identities (LGBTQ+) and underrepresented in medicine (URiM) trainee parents, who have been underrepresented in previous research on trainee parents and face barriers that make it harder to balance family life and training. LGBTQ+ parents often have fewer benefits and unique challenges, such as limited access to parental leave and more frequent use of assisted reproductive technology, while URiM parents face compounded challenges from the intersectionality of their identities.

The expected outcome of this project is the development of a structured, scalable coaching program that reduces burnout in childbearing trainees by integrating one-on-one coaching with community-building and group support. This program will have a significant positive impact on the clinical learning environment by enhancing its diversity, equity, and belonging while improving the well-being of a vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. English fluency and literacy
3. Resident or fellow level MD or DO trainee
4. Pregnant or up to 3 months post-partum

Exclusion Criteria:

1. Unable to provide consent.
2. Unable to complete electronic surveys and video calls.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Burnout | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  8-item Emotional Exhaustion (EE) and Depersonalization (DP) subscales in the Stanford Professional Fulfillment Index (SPFI). Higher scores are associated with more feelings of burnout while lower scores are associated with lower levels of burnout.

SECONDARY OUTCOMES:
Burnout | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  Six item abbreviated version of the Maslach Burnout Inventory, including the Emotional Exhaustion (EE) and Depersonalization (DP) subscales. Higher scores are associated with higher levels of burnout while lower scores are associated with lower levels of burnout.
Professional fulfillment | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  Four item Stanford Professional Fulfillment Index subscale. Higher scores are associated with higher measures of professional fulfillment, and lower scores are associated with lower levels of professional fulfillment.
Imposter Phenomenon | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  20-question Clance Imposter Phenomenon Scale. Imposter phenomenon - associated with work-life integration challenges, burnout, and low professional fulfillment - is more common in high-achieving women during times of life transition and causes self-doubt despite objective evidence of achievement. Higher scores are associated with high feelings of imposter phenomenon and low scores are associated with less imposter phenomenon.
Self-valuation | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  Four item Clinician Self-Valuation scale. Low self-valuation - associated with burnout - is more common in women. It includes a harsh response to perceived personal shortcomings and deferral of personal needs to meet others' needs to meet others' needs. High scores are associated with low self-valuation while low scores are associated with high self-valuation.
Self-efficacy | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  Eight item New Generalized Self-Efficacy Scale. Self-efficacy is an individuals' perceived ability to perform across challenges, associated with lower levels of emotional exhaustion. High scores are associated with high levels of self-efficacy, low scores are associated with low levels of self-efficacy.
Resilience | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  Two item Connor Davidson Resilience Scale. Resilience - negatively correlated with physician burnout - includes adaptability to stress, a growth mindset, and enhanced social support, and improves with professional coaching. High scores are associated with high levels of resilience while low scores are associated with low levels of resilience.
Quality of life (QoL) | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  single-item validated linear analogue self-assessment
Impact of Work on Personal Relationships | Measured in survey data at 3 time points: Enrollment, month 4 and month 7 of study.
  Four-item Stanford Professional Fulfillment Index - Impostor Work Performance Relations (IWPR) Scale. Higher scores are associated with greater feelings of social isolation, burnout, and increased patient complaints.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlick CJR, Ellis RJ, Etkin CD, Greenberg CC, Greenberg JA, Turner PL, Buyske J, Hoyt DB, Nasca TJ, Bilimoria KY, Hu YY. Experiences of Gender Discrimination and Sexual Harassment Among Residents in General Surgery Programs Across the US. JAMA Surg. 2021 Oct 1;156(10):942-952. doi: 10.1001/jamasurg.2021.3195. PMID 34319377
- [Background] Rangel EL, Smink DS, Castillo-Angeles M, Kwakye G, Changala M, Haider AH, Doherty GM. Pregnancy and Motherhood During Surgical Training. JAMA Surg. 2018 Jul 1;153(7):644-652. doi: 10.1001/jamasurg.2018.0153. PMID 29562068
- [Background] Li RD, Janczewski LM, Eng JS, Foote DC, Wu C, Johnson JK, Easter SR, Kim E, Buyske J, Turner PL, Nasca TJ, Bilimoria KY, Hu YY, Rangel EL. Pregnancy and Parenthood Among US Surgical Residents. JAMA Surg. 2024 Oct 1;159(10):1127-1137. doi: 10.1001/jamasurg.2024.2399. PMID 39018050
- [Background] Rowe SG, Stewart MT, Van Horne S, Pierre C, Wang H, Manukyan M, Bair-Merritt M, Lee-Parritz A, Rowe MP, Shanafelt T, Trockel M. Mistreatment Experiences, Protective Workplace Systems, and Occupational Distress in Physicians. JAMA Netw Open. 2022 May 2;5(5):e2210768. doi: 10.1001/jamanetworkopen.2022.10768. PMID 35522279
- [Background] National Academies of Sciences, Engineering, and Medicine; National Academy of Medicine; Committee on Systems Approaches to Improve Patient Care by Supporting Clinician Well-Being. Taking Action Against Clinician Burnout: A Systems Approach to Professional Well-Being. Washington (DC): National Academies Press (US); 2019 Oct 23. Available from http://www.ncbi.nlm.nih.gov/books/NBK552618/ PMID 31940160
- [Background] Sullivan MC, Bucholz EM, Yeo H, Roman SA, Bell RH, Sosa JA. "Join the club": effect of resident and attending social interactions on overall satisfaction among 4390 general surgery residents. Arch Surg. 2012 May;147(5):408-14. doi: 10.1001/archsurg.2012.27. PMID 22785631
- [Background] Dyrbye LN, Shanafelt TD, Gill PR, Satele DV, West CP. Effect of a Professional Coaching Intervention on the Well-being and Distress of Physicians: A Pilot Randomized Clinical Trial. JAMA Intern Med. 2019 Oct 1;179(10):1406-1414. doi: 10.1001/jamainternmed.2019.2425. PMID 31380892
- [Background] Palamara K, McKinley SK, Chu JT, Merrill AL, Yu L, Parangi S, Makowski MS, Park YS, Donelan K, Stein SL. Impact of a Virtual Professional Development Coaching Program on the Professional Fulfillment and Well-Being of Women Surgery Residents: A Randomized Controlled Trial. Ann Surg. 2023 Feb 1;277(2):188-195. doi: 10.1097/SLA.0000000000005562. Epub 2022 Jun 29. PMID 35766397
- [Background] Fainstad T, Mann A, Suresh K, Shah P, Dieujuste N, Thurmon K, Jones CD. Effect of a Novel Online Group-Coaching Program to Reduce Burnout in Female Resident Physicians: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2210752. doi: 10.1001/jamanetworkopen.2022.10752. PMID 35522281
- [Background] Lyu HG, Davids JS, Scully RE, Melnitchouk N. Association of Domestic Responsibilities With Career Satisfaction for Physician Mothers in Procedural vs Nonprocedural Fields. JAMA Surg. 2019 Aug 1;154(8):689-695. doi: 10.1001/jamasurg.2019.0529. PMID 30969336